CLINICAL TRIAL: NCT03942042
Title: A Multicenter, Open-Label, Post Marketing Clinical Trial to Evaluate the Efficacy And Safety Of Ixekizumab in Patients With Generalized Pustular Psoriasis and Erythrodermic Psoriasis
Brief Title: A Study of Ixekizumab (LY2439821) in Participants in Japan With Generalized Pustular Psoriasis and Erythrodermic Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17154; I1F-JE-RHCV (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Generalized Pustular Psoriasis; Erythrodermic Psoriasis
Keywords: Generalized Pustular Psoriasis (GPP); Erythrodermic Psoriasis (EP); Japan
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ixekizumab (Experimental): Induction Dosing Period:
  Participants received 160 milligrams (mg) ixekizumab subcutaneously (SC) as 2 injections at Week 0 followed by 80 mg ixekizumab SC as 1 injection at Week 2, 4, 6, 8 and 10.
  Maintenance Dosing Period:
  Participants with Global Improvement Score (GIS) = 1 at Week 12 are responders who will complete the study.
  Participants who are inadequate responders (GIS ≥2 at Week 12 and based on the investigators' discretion) will be administered 80 mg ixekizumab SC as 1 injection at Week 12, 14, 16, and 18 or until they achieve a GIS score of 1.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
The reason for this study is to see if the study drug ixekizumab is safe and effective in participants with generalized pustular psoriasis and erythrodermic psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Present with GPP or EP based on an investigator-confirmed diagnosis and meet the associated criteria

  * GPP: Meet the criteria for GPP set by Ministry of Health, Labour and Welfare (MHLW) at screening and baseline regardless of IL-36 mutation status.
  * EP: Diagnosed to have BSA ≥80% involvement (with inflammatory erythema) at screening and baseline.
* Candidates for phototherapy and/or systemic therapy
* Men must agree to use a reliable method of birth control during the study
* Women must agree to use birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* History of drug-induced psoriasis
* Concurrent or recent use of any biologic agent
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to enrollment and during the study
* Have previously received ixekizumab
* Serious disorder or illness other than psoriasis
* Serious infection within the last 12 weeks
* Breastfeeding or nursing (lactating) women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Japan (7):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Jikei University School of Medicine, Minato-Ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Osaka City University Medical School Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Morita A, Okubo Y, Morisaki Y, Torisu-Itakura H, Umezawa Y. Ixekizumab 80 mg Every 2 Weeks Treatment Beyond Week 12 for Japanese Patients with Generalized Pustular Psoriasis and Erythrodermic Psoriasis. Dermatol Ther (Heidelb). 2022 Feb;12(2):481-494. doi: 10.1007/s13555-021-00666-x. Epub 2021 Dec 29. PMID 34967916

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixekizumab - Generalized Pustular Psoriasis (GPP): Induction Dosing Period:
  Participants received 160 milligrams (mg) ixekizumab subcutaneously (SC) as 2 injections at Week 0 followed by 80 mg ixekizumab SC as 1 injection at Week 2, 4, 6, 8 and 10.
  Maintenance Dosing Period:
  Participants with Global Improvement Score (GIS) = 1 at Week 12 are responders who will complete the study.
  Participants who are inadequate responders (GIS ≥2 at Week 12 and based on the investigators' discretion) will be administered 80 mg ixekizumab SC as 1 injection at Week 12, 14, 16, and 18 or until they achieve a GIS score of 1.
- Ixekizumab - Erythrodermic Psoriasis (EP): Induction Dosing Period:
  Participants received 160 mg ixekizumab SC as 2 injections at Week 0 followed by 80 mg ixekizumab SC as 1 injection at Week 2, 4, 6, 8 and 10.
  Maintenance Dosing Period:
  Participants with Global Improvement Score (GIS) = 1 at Week 12 are responders who will complete the study.
  Participants who are inadequate responders (GIS ≥2 at Week 12 and based on the investigators' discretion) will be administered 80 mg ixekizumab SC as 1 injection at Week 12, 14, 16, and 18 or until they achieve a GIS score of 1.
Period: Induction Dosing Period (12 Weeks)
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Started | 7 | 5
Received at Least One Dose of Study Drug | 7 | 5
Participants With GIS=1 at Week 12 | 4 | 0
Participants Who Completed Week 12 With GIS >= 2 | 2 | 4
Completed | 6 | 4
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 1 | 0
Period: Maintenance Dosing Period (8 Weeks)
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Started | 2 (Only participants with GIS ≥2 at Week 12 and based on investigators' discretion continued to maintenance dosing period.) | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Ixekizumab - Generalized Pustular Psoriasis (GPP); Ixekizumab - Erythrodermic Psoriasis (EP): Induction Dosing Period:
  Participants received 160 mg ixekizumab SC as 2 injections at Week 0 followed by 80 mg ixekizumab SC as 1 injection at Week 2, 4, 6, 8 and 10.
  Maintenance Dosing Period:
  Participants with Global Improvement Score (GIS) = 1 at Week 12 are responders who will complete the study.
  Participants who are inadequate responders (GIS ≥2 at Week 12 and based on the investigators' discretion) will be administered 80 mg ixekizumab SC as 1 injection at Week 12, 14, 16, and 18 or until they achieve a GIS score of 1.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP) | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (19.10) | 42.2 (14.39) | 43.8 (16.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Dosing Period: Number of Participants Who Improved Global Improvement Score (GIS) at Least 1 Point From Week 12 Through Week 20 and With ≤2 of GIS
Description: GIS was assessed in the 4 grades by comparing the psoriatic findings: (1) resolved, (2) improved, (3) unchanged, or (4) worsened. The global improvement score was assessed based on the comparison of the psoriatic findings, Static Physician Global Assessment (sPGA), Psoriasis Area and Severity Index (PASI) score, and other evaluations with those at the baseline.
Time Frame: Week 12 through Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Ixekizumab - Generalized Pustular Psoriasis (GPP); Ixekizumab - Erythrodermic Psoriasis (EP): Maintenance Dosing Period:
  Participants with Global Improvement Score (GIS) = 1 at Week 12 are responders who will complete the study.
  Participants who are inadequate responders (GIS ≥2 at Week 12 and based on the investigators' discretion) will be administered 80 mg ixekizumab SC as 1 injection at Week 12, 14, 16, and 18 or until they achieve a GIS score of 1.
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 1 | 0

2. Secondary Outcome: Maintenance Dosing Period: Number of Participants With GIS Grade 1: Resolved
Description: as for outcome 1
Time Frame: Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 1 | 0

3. Secondary Outcome: Maintenance Dosing Period: Number of Participants With GIS Grade 2: Improved
Description: as for outcome 1
Time Frame: Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 1 | 4

4. Secondary Outcome: Maintenance Dosing Period: Number of Participants With GIS Grade 3: Unchanged
Description: as for outcome 1
Time Frame: Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

5. Secondary Outcome: Maintenance Dosing Period: Number of Participants With GIS Grade 4: Worsened
Description: as for outcome 1
Time Frame: Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

6. Secondary Outcome: Maintenance Dosing Period: Number of Participants Who Achieved Static Physician Global Assessment (sPGA) of (0, 1)
Description: The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA assessed as either 0 or 1 represents a clinically meaningful response of minimal plaque severity or complete resolution of psoriasis.
Time Frame: Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 2 | 1

7. Secondary Outcome: Maintenance Dosing Period: Number of Participants Who Achieved at Least a 75% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score (PASI 75) Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score (PASI 75)
Description: PASI combines assessments of the extent of body surface involvement in 4 regions (head & neck(h), trunk(t), arms(u), legs(l)) & severity of scaling (S), redness (R), & plaque induration/infiltration (thickness, T) in each region. Severity is rated for each index (R, S, T) on a 0-4 scale (0 for no involvement up to 4 for severe involvement): 0 = none, 1 = slight, 2 = mild, 3 = moderate, 4 = severe Fraction of total body surface area (BSA) affected is graded on a 0-6 scale (0 for no involvement to 6 for 90% - 100% involvement): 0 = 0% (clear), 1 = >0% to <10%, 2 = 10% to <30%, 3 = 30% to <50%, 4 = 50% to <70%, 5 = 70% to 90%, 6 = 90% to 100%.
  Overall score ranges from 0 (no psoriasis) to 72 (most severe disease).
Time Frame: Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 2 | 3

8. Secondary Outcome: Maintenance Dosing Period: Change From Baseline in Psoriasis Scalp Severity Index (PSSI) in Participants With Scalp Involvement at Baseline
Description: The scalp was assessed for erythema (redness), induration (hardness), and desquamation (shedding of skin) and percentage of area affected as follows:
  Erythema, Induration and Desquamation:
  0 = Absent
  1. = Slight
  2. = Moderate
  3. = Severe
  4. = Severest Possible
  Percent of Scalp Involved:
  1. = <10%
  2. = 10% - 29%
  3. = 30% - 49%
  4. = 50% - 69%
  5. = 70% - 89%
  6. = 90% - 100%
  The PSSI score is a composite score derived from the sum of the scores for erythema, induration and desquamation multiplied by the score for the extent of scalp area involved (percent of scalp involved). The range is 0 (no psoriasis) to 72 (Most severe Disease).
Time Frame: Baseline, Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug who had Scalp Involvement at Baseline.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 1 | 4
units on a scale | -9.0 [-9.0 to -9.0] | -25.5 [-46.0 to -15.0]

9. Secondary Outcome: Maintenance Dosing Period: Change From Baseline in Percent of Body Surface Area (BSA) Involvement of Psoriasis Body Surface Area (BSA) Involvement of Psoriasis
Description: Percentage involvement of psoriasis on each participants body surface area was assessed by the investigator on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand (including palm, fingers and thumb).
Time Frame: Baseline, Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
units on a scale | -44.5 [-64 to -25] | -61.3 [-89 to -7]

10. Secondary Outcome: Maintenance Dosing Period: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI is a simple, patient-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all", "a little","a lot", and "very much", with corresponding scores of 0, 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (the higher the score, the more quality of life is impaired) and a 5-point change from baseline is considered clinically relevant (Basra et al. 2008).
Time Frame: Baseline, Week 20
Population: Maintenance Dosing Period: All randomized participants who received at least one dose of study drug.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
score on a scale | -4.0 [-9 to 1] | -6.5 [-18 to -1]

11. Secondary Outcome: Maintenance Dosing Period: Number of Participants Who Developed Treatment-Emergent Anti-Ixekizumab Antibodies (TE-ADA)
Description: Number of participants who developed treatment-emergent anti-ixekizumab antibodies (TE-ADA) was summarized by treatment group.
Time Frame: Week 20
Population: Maintenance Dosing Period: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

12. Secondary Outcome: Maintenance Dosing Period: Number of Participants Who Developed Neutralizing Anti-Ixekizumab Antibody (NAb)
Description: Number of participants who developed neutralizing Anti-Ixekizumab antibody (NAb) was summarized by treatment group.
Time Frame: Week 20
Population: Maintenance Dosing Period: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP) | Ixekizumab - Erythrodermic Psoriasis (EP)
Number analyzed (Participants) | 2 | 4
Participants | 0 | 0

13. Secondary Outcome: Generalized Pustular Psoriasis (GPP) Only: Change From Baseline on Generalized Pustular Psoriasis Severity Index
Description: GPP Severity Index was evaluated only for participants with pustular psoriasis at screening and at baseline. This is a composite score derived from the sum of scores for assessment of dermal symptoms, systemic symptoms, and laboratory findings (range, 0 to 17, with 17 representing severe symptoms). Skin symptoms were assessed by the score with the area of erythema (on a 0 to 3 scale), area of confluent pustules (on a 0 to 3 scale), and are of skin edema (on a 0 to 3 scale). The total score will be assessed (range, 0 to 9, with 9 representing severe symptoms). Systemic symptoms and laboratory findings were assessed by the score with fever (on a 0 to 2 scale), white blood cell (on a 0 to -2 scale), C-reactive protein (on a 0 to 2 scale) and Albumin (on a 0 to 2 scale). The total score will be assessed (range, 0 to 8, with 8 representing severe symptoms).
Time Frame: Baseline, Week 20
Population: Maintenance Dosing Period: All participants who received at least one dose of study drug in GPP arm.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ixekizumab - Generalized Pustular Psoriasis (GPP)
Number analyzed (Participants) | 2
units on a scale | -2.5 [-4 to -1]

ADVERSE EVENTS:
Time Frame: Baseline Up To 20 Weeks
Description: All participants who received at least one dose of study drug.
Groups:
- Ixekizumab GPP-Induction Dosing Period; Ixekizumab EP-Induction Dosing Period: Induction Dosing Period:
  Participants received 160 mg ixekizumab SC as 2 injections at Week 0 followed by 80 mg ixekizumab SC as 1 injection at Week 2, 4, 6, 8 and 10.
- Ixekizumab GPP-Combined Induction and Maintenance Periods; Ixekizumab EP-Combined Induction and Maintenance Periods: Maintenance Dosing Period:
  Participants with Global Improvement Score (GIS) = 1 at Week 12 are responders who will complete the study.
  Participants who are inadequate responders (GIS ≥2 at Week 12 and based on the investigators' discretion) will be administered 80 mg ixekizumab SC as 1 injection at Week 12, 14, 16, and 18 or until they achieve a GIS score of 1.
Arm/Group | Ixekizumab GPP-Induction Dosing Period | Ixekizumab EP-Induction Dosing Period | Ixekizumab GPP-Combined Induction and Maintenance Periods | Ixekizumab EP-Combined Induction and Maintenance Periods
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/5 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 4/7 | 2/5 | 1/2 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab GPP-Induction Dosing Period (N=7) | Ixekizumab EP-Induction Dosing Period (N=5) | Ixekizumab GPP-Combined Induction and Maintenance Periods (N=2) | Ixekizumab EP-Combined Induction and Maintenance Periods (N=4)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab GPP-Induction Dosing Period (N=7) | Ixekizumab EP-Induction Dosing Period (N=5) | Ixekizumab GPP-Combined Induction and Maintenance Periods (N=2) | Ixekizumab EP-Combined Induction and Maintenance Periods (N=4)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT03942042/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03942042/SAP_001.pdf